CLINICAL TRIAL: NCT01643577
Title: Acupuncture Treatment for Gastroparesis: a Pilot Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Linda A. Lee, MD, Principal Investivator, Associate Professor of Medicine, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NA_00044436
Record Dates: First submitted 2012-06-26; First posted 2012-07-18 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Gastroparesis; Nausea; Vomiting; Abdominal Pain
Keywords: Idiopathic; gastroparesis; delayed gastric emptying; nausea; vomiting; abdominal pain; bloating
MeSH Terms: conditions — Gastroparesis; Nausea; Vomiting; Abdominal Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acupuncture protocol for gastroparesis (Active Comparator): Patients randomized to this arm will receive an acupuncture protocol that with points designed to treat gastroparesis
  Interventions: Procedure: Acupuncture for gastroparesis
- Acupuncture for musculoskeletal pain (Placebo Comparator): Patients randomized to this arm will receive acupuncture therapy consisting of points designed to treat musculoskeletal pain.
  Interventions: Procedure: Acupuncture for musculoskeletal pain

INTERVENTIONS:
Procedure: Acupuncture for gastroparesis — A series of acupuncture points selected for the treatment of gastroparesis will be used at each of the 10 acupuncture sessions
  Arms: Acupuncture protocol for gastroparesis
Procedure: Acupuncture for musculoskeletal pain — Acupuncture points selected for the treatment of musculoskeletal pain will be used during each of the 10 acupuncture sessions
  Arms: Acupuncture for musculoskeletal pain

SUMMARY:
Gastroparesis is a disorder characterized by delayed gastric emptying leading to symptoms of nausea, vomiting, bloating, and abdominal pain. A common cause is diabetes but even more often it occurs in otherwise healthy individuals. The symptoms of gastroparesis can significantly alter a patient's quality of life. Current therapies are limited. In this study, the investigators seek to determine if twice weekly acupuncture treatments can improve symptoms of gastroparesis.

DETAILED DESCRIPTION:
Gastroparesis is a disorder characterized by delayed gastric emptying leading to symptoms of nausea, vomiting, bloating, and abdominal pain. A common cause is diabetes but often it occurs in otherwise healthy individuals in whom the disorder is said to be idiopathic. The symptoms of gastroparesis can significantly alter a patient's quality of life and may result in absenteeism or frequent ER visits and hospitalizations for dehydration caused by intractable nausea and vomiting.

Current treatment for gastroparesis includes dietary and lifestyle modifications, tight glycemic control in diabetics, and supportive care for symptoms, like anti-emetics for nausea. Prokinetic therapies to enhance gastric emptying such as metoclopramide, domperidone, and erythromycin have varying degrees of effect. Unfortunately they are often limited by side effects. Metoclopramide, the only pharmacologic agent that is FDA approved for the treatment of gastroparesis, in particular crosses the blood brain barrier and may cause CNS side effects, reported to be 10-25% of the time. The most rare but most worrisome adverse reaction is tardive dyskinesia associated with prolonged use of metoclopramide, prompting the FDA to label it with a blackbox warning. Use of erythromycin is limited to acute flares, as prolonged use causes tachyphylaxis. Finally, domperidone may have equal efficacy as metoclopramide and is available in 58 countries. However, it is not FDA approved in the US but can be obtained with an Investigational New Drug Application. Given these constraints, novel therapies to improve symptoms are needed.

Preliminary studies from Asia and the US have shown a potential role for acupuncture in improving gastroparetic symptoms and gastric motility in diabetic and non-diabetic patients. It is our plan to expand on the available research by using validated instruments to measure changes in severity of symptoms and quality of life, incorporating randomization and blinding, and correcting for possible placebo effect.

Our hypothesis is that twice weekly acupuncture treatments can improve symptoms of gastroparesis with an effect that lasts beyond the last treatment date without inducing side-effects. We also hypothesize that gastric emptying may improve compared to baseline values. This is a pilot study of 20 gastroparetic patients who will be randomized to standard medical therapy + acupuncture designed to treat gastroparesis vs. standard medical therapy + acupuncture designed to treat unrelated musculoskeletal and arthralgia complaints.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be at least 18 years old and able to provide informed consent.
* Participants will have symptoms of idiopathic gastroparesis for at least 6 months duration prior to enrollment with documented abnormal solid phase gastric emptying scintigraphy

Exclusion Criteria:

* Gastroparesis due to: diabetes, medication (e.g. post-chemotherapy), iatrogenic post-surgical gastroparesis, and severe neurologic conditions such as Parkinson's disease known to be associated with gastroparesis.
* An active eating disorder,
* Participants currently lactating, or preparing to conceive will also be excluded.
* A history of inflammatory bowel disease
* Known bowel obstruction, or strictures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Symptomatic improvement using GCSI | 10 weeks
  To determine whether acupuncture treatment designed to treat gastroparesis significantly improves symptoms of gastroparesis measured by the Gastroparesis cardinal symptoms index (GCSI)

SECONDARY OUTCOMES:
Gastric emptying time | 5 weeks
  To determine whether acupuncture treatment designed to treat gastroparesis significantly improves gastric emptying measured by the Smart Pill
Small bowel and colonic transit time | 5 weeks
  To determine whether acupuncture treatment designed to treat gastroparesis significantly alters small bowel and colonic motility using Smart Pill

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Integrative Medicine & Digestive Center, Lutherville, Maryland, United States